CLINICAL TRIAL: NCT01613443
Title: Time-dependent ex Vivo Influence of Rivaroxaban on Point-of-care Devices
Brief Title: Ex-vivo Effect of New Oral Anticoagulants on Point-of-care Devices
Status: Completed | Type: Observational
Sponsor: Cardioangiologisches Centrum Bethanien (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. E. Lindhoff-Last, Prof. Dr. med. Lindhoff-Last, Cardioangiologisches Centrum Bethanien
Other Study IDs: POCT-NOAC
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Effect of NOAC on POCT
Keywords: Dabigatran, Rivaroxaban, Point of Care-testing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Control: Healthy volunteers without medication
- Phenprocoumon: Patients receiving Marcumar having target INR 2-3
- Dabigatran: Patients receiving therapeutic dosis of Pradaxa
- Rivaroxaban: Patients receiving therapeutic dosis of Xarelto

SUMMARY:
Concentration determinations of anticoagulants require plasma instead of whole blood, and results are not immediately available to clinicians. Monitoring anticoagulants concentration along with bedside methods may provide an alternative guide for administration of the NOAC.

The purpose of this investigation is to compare bedside coagulation assays in whole blood with plasma concentrations of the new oral anticoagulants (NOAC) in patients treated with therapeutic dosis of NOAC.

DETAILED DESCRIPTION:
This open-label study will be performed by ex vivo investigations. Patients receiving the NOAC as dabigatran or rivaroxaban in therapeutic doses are recruited and informed consent of two blood sampling times will be obtained in correlation to the time of drug intake (two and 24 hours after drug intake). The bedside measurements will be performed and compared directly with the concentrations determined by plasma concentration assays. These investigations will be performed at the department of Angiology at the university hospital Frankfurt.

ELIGIBILITY:
The indication for the use of NOAC is provided by the attending physician. The criteria for inclusion and exclusion criteria for the use of the new oral anticoagulants must meet appropriate eligibility criteria and the clinical guidelines that are described in the SOPs.

Patients treated with dabigatran 2x150mg / d for the prevention of stroke and systemic embolism in non-valvular atrial fibrillation are included.

Moreover, patients treated with rivaroxaban 20 mg / d for DVT prophylaxis and treatment of recurrent DVT or PE are included.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients indicated for NOAC-therapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-06; Primary Completion 2013-05 (Actual); Study Completion 2013-08 (Actual)

REFERENCES:
- [Result] Mani H, Herth N, Kasper A, Wendt T, Schuettfort G, Weil Y, Pfeilschifter W, Linnemann B, Herrmann E, Lindhoff-Last E. Point-of-care coagulation testing for assessment of the pharmacodynamic anticoagulant effect of direct oral anticoagulant. Ther Drug Monit. 2014 Oct;36(5):624-31. doi: 10.1097/FTD.0000000000000064. PMID 24577124